CLINICAL TRIAL: NCT06539637
Title: Ketorolac Levels in Vitreous and Aqueous Samples From Patients Undergoing Combined Cataract and Pars Plana Vitrectomy Surgeries With and Without Intracameral Phenylephrine 1.0% / Ketorolac 0.3%
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: DHS Consulting (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00068701
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Phenylephrine; Ketorolac; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- OMIDRIA (Active Comparator): OMIDRIA is a combination product containing 10.16 mg/mL (1% w/v) of phenylephrine and 2.88 mg/mL (0.3% w/v) of ketorolac in a single-patient-use vial. Once the 4mL of OMIDRIA is diluted in 500 mL of ophthalmic irrigation solution, the resulting solution is intended to be used as needed during cataract surgery or intraocular lens replacement.
  Interventions: Combination Product: OMIDRIA (*Registered Product) {10.16 mg/mL (1% w/v) of phenylephrine and 2.88 mg/mL (0.3% w/v) of ketorolac}
- Topical Ketorolac (Active Comparator): Topical ketorolac tromethamine 0.5% is a nonsteroidal anti-inflammatory drug. It is FDA-approved for the treatment of inflammation following cataract surgery and relief of ocular itching due to seasonal allergic conjunctivitis.
  Interventions: Other: Ketorolac Tromethamine {TORADOL} (0.5%) - Topical Eyedrop

INTERVENTIONS:
Combination Product: OMIDRIA (*Registered Product) {10.16 mg/mL (1% w/v) of phenylephrine and 2.88 mg/mL (0.3% w/v) of ketorolac} — 10.16 mg/mL (1% w/v) of phenylephrine {Generic Name: Biorphen} (Adrenergic Receptor Agonist) and 2.88 mg/mL (0.3% w/v) of ketorolac {Generic Name: TORADOL} (Nonsteroidal Anti-inflammatory) - via intracameral delivery
  Arms: OMIDRIA
Other: Ketorolac Tromethamine {TORADOL} (0.5%) - Topical Eyedrop — Topical ketorolac tromethamine {TORADOL, Nonsteroidal Anti-inflammatory} (0.5%) administered 4 times daily for the 3 days leading up to surgery. The last drop is to be given at least 2 hours prior to surgery.
  Arms: Topical Ketorolac

SUMMARY:
This is a clinical trial evaluating Ketorolac levels in vitreous and aqueous humor samples from patients undergoing combined cataract and pars plana vitrectomy surgeries with and without intracameral phenylephrine 1.0% / ketorolac 0.3% (OMIDRIA). Patients not receiving intracameral OMIDRIA will receive topical ketorolac prior to cataract surgery/pars plana vitrectomy.

DETAILED DESCRIPTION:
Cataract surgery can result in intra- and postoperative inflammation. Various strategies are employed to prevent and combat this inflammatory reaction, including preoperative topical NSAIDs, intraoperative NSAIDs or steroids, and postoperative topical NSAIDs and/or steroids. The only FDA-approved NSAID for intraoperative use is the ketorolac component of OMIDRIA® (Rayner Surgical, Bellevue, WA, USA).

Animal studies have assessed the concentration of ketorolac in the vitreous and demonstrated therapeutic levels out to 10 hours postoperatively. There is no human data for ketorolac levels in the vitreous following intracameral administration of OMIDRIA at the time of cataract surgery.

This study will enroll approximately 10-20 patients undergoing combined cataract surgery immediately followed by pars plana vitrectomy. Aqueous and vitreous samples will be taken intraoperatively and sent to an independent lab for analysis of ketorolac concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Undergoing cataract surgery immediately followed by pars plana vitrectomy
3. Diagnosed preoperatively with a structural pathology requiring vitrectomy (e.g., epiretinal membrane, macular hole, and symptomatic vitreous floaters)
4. Willing and able to comply with all study procedures
5. Male or female, aged ≥ 18 years

Exclusion Criteria:

1. Age < 18
2. Participating in another clinical trial
3. Patients undergoing cataract surgery or pars plana vitrectomy alone (not a combined procedure)
4. Previous vitrectomy
5. Complications at the time of cataract surgery
6. A tear in the posterior capsule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Concentration of ketorolac in the vitreous humor | The day of surgery
  Vitreous samples taken from vitrectomy at the beginning of the procedure for all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donnenfeld, MD, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (1):
- Ophthalmic Consultants of Long Island, Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No